CLINICAL TRIAL: NCT00997334
Title: First-Line Erlotinib Therapy and the Subsequent Development of Mechanisms of Secondary Resistance in Patients With Non-Small Cell Lung Cancer and Known Sensitizing EGFR Mutations
Brief Title: Erlotinib Therapy and Subsequent Development of Mechanisms of Secondary Resistance in Patients With NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David M. Jackman, MD (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David M. Jackman, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-210; NE_OSI4590s (Other: Genentech/Roche)
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: erlotinib; EGFR mutation; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental): Erlotinib was given at a dose of 150mg orally once per day for 28 days (+/- 3 days); Patients are treated until disease progression or until unaccepted drug toxicity.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib
  Other Names: Tarceva

SUMMARY:
Erlotinib is a drug which targets non small cell lung cancer with a genetic change (mutation) in the epidermal growth factor receptor (EGFR). This drug has been used in other cancer research studies and information from those studies suggests that Erlotinib can control the growth of these cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

-To prospectively assess the frequency of different genetic mechanisms of secondary resistance in patients' tumors during treatment with erlotinib (e.g., T790M mutations, MET amplification).

* Correlate these genetic changes with patient demographic data and clinical outcomes (time to progression, survival, sites of recurrence/progression).
* Search for novel mechanisms of acquired resistance to erlotinib.
* Identify whether these genetic changes are present at low levels in initial pretreatment tumor specimens.

SECONDARY OBJECTIVE(S)

1. To measure the steady-state plasma concentrations of erlotinib during the course of patients' treatment.

   * Determine if the development and/or resolution of skin toxicity is related to plasma erlotinib concentrations.
   * Determine if the development of disease progression while on erlotinib is correlated with declines in plasma erlotinib concentrations.
   * Assess the plasma levels in patients whose smoking status has been biochemically verified to determine if smoking is associated with lower erlotinib plasma concentration.
2. To analyze from both free plasma DNA and DNA from circulating tumor cells of erlotinib-treated patients for the original sensitizing EGFR mutations and genetic changes associated with secondary resistance.
3. To measure clinical outcomes in patients with known sensitizing mutations in their tumor EGFR when treated with first-line erlotinib.

   * Response rate
   * Time to progression
   * Median overall survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer, stage IV or IIIB with a malignant pleural or pericardial effusion. Patients with stage I or II non-small cell lung cancer who have undergone surgical resection but who subsequently relapse with metastatic disease or a malignant pleural effusion are also eligible.
* Documentation of a sensitizing mutation of the epidermal growth factor receptor. In addition, there must be a sufficient tissue for analysis of KRAS (the oncogene from the Kirsten rat sarcoma virus) mutations and MET amplification.
* At least one measurable or evaluable site of disease as defined by revised RECIST (version 1.1) criteria.
* 18 years of age or older
* No more than one prior systemic therapy regimen for advanced non-small cell lung cancer. Chemotherapy delivered as part of concurrent chemoradiation will also count as a prior systemic therapy regimen. Adjuvant therapy for resected NSCLC will not count towards this total as long as it was completed at least 6 months prior to enrollment and did not include therapy with an EGFR-targeted agent. Adjuvant therapy completed less than 6 months prior to the time of screening will count as a prior regimen.
* 3 or more weeks since prior major surgery
* 2 or more weeks since prior radiation
* ECOG performance status 0-1
* Life expectancy > 8 weeks
* Adequate hematologic, renal, and hepatic function
* Willingness to undergo repeat tumor biopsy at the time of disease progression.

Exclusion Criteria:

* Untreated and/or uncontrolled central nervous system metastases. Patients with prior brain metastases must have had definitive treatment (radiation or surgery) and must be clinically stable off steroids for at least 1 week prior to enrollment.
* More than one prior systemic chemotherapy for advanced non-small cell lung cancer. , Chemotherapy delivered as part of concurrent chemoradiation will also count as a prior systemic therapy regimen. Adjuvant therapy for resected NSCLC willnot count towards this total as long as it was completed at least 6 months prior to enrollment and did not include therapy with an EGFR-targeted agent. Adjuvant therapy completed less than 6 months prior to the time of screening will count as a prior regimen.
* Prior exposure to erlotinib or other treatments targeting the HER family axis.
* Active malignancies within the past 3 years, except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Any process that compromises the ability to swallow and/or absorb oral medication.
* Incomplete healing from previous surgery
* A history of any of the following autoimmune skin disorders: Sjogren's syndrome, scleroderma, dermatomyositis, and systemic lupus erythematosus.
* Significant medical history or unstable medical conditions.
* Concurrent use of warfarin. Patients must be off warfarin for at least one week prior to initiation of erlotinib. Other non-warfarin anticoagulants are permitted.
* Patients who require ongoing concomitant use of one of the strong inhibitors/inducers of CYP3A4.
* Pregnant or breastfeeding. Women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jackman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Redig AJ, Costa DB, Taibi M, Boucher D, Johnson BE, Janne PA, Jackman DM. Prospective Study of Repeated Biopsy Feasibility and Acquired Resistance at Disease Progression in Patients With Advanced EGFR Mutant Lung Cancer Treated With Erlotinib in a Phase 2 Trial. JAMA Oncol. 2016 Sep 1;2(9):1240-2. doi: 10.1001/jamaoncol.2016.1304. No abstract available. PMID 27387964

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study activated December 2009. Patients enrolled from February 2010 - January 2015
Period: Overall Study
Arm/Group | Erlotinib
Started | 60
Eligible for Repeat Biopsy | 44 (Patients who experience disease progression on treatment were eligible for repeat biopsy)
Evaluable | 35 (Patients with tissue available for re-biopsy at time of progression)
Completed | 35
Not Completed | 25
Not completed — still on therapy | 12
Not completed — Adverse Event | 3
Not completed — Patient non-compliance | 1
Not completed — Withdrawal by Subject | 3
Not completed — Death | 2
Not completed — Urgent Palliative Care | 2
Not completed — No lesion amenable | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Population: The analysis data is comprised of all treated patients
Groups:
- Erlotinib: Patients receive standard dose of erlotinib 150mg daily with cycle length of 28 days; Patients are treated until disease progression or until unaccepted drug toxicity.
Arm/Group | Erlotinib
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 60 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60
Smoking Status [Count of Participants; unit: Participants]
  Never-Smoker | 34
  Smoker | 26

OUTCOME MEASURES:

1. Primary Outcome: Resistance Mechanism
Description: Participants were classified into 4 potential resistant mechanism groups (4 genetic/ 1 histologic) based on evaluation of rebiopsy tissue: EGFR mutations (T790M mutation, exon 20 insertion), KRAS mutations, MET amplification or small-cell lung cancer (SCLC) transform using established methods.
Time Frame: Participants were evaluated for incidence of genetic mechanisms of secondary resistance at time of disease progression at which point participants stopped treatment. Progression follow up was up to 3 years in this study cohort.
Population: The analysis dataset is comprised of all evaluable patients.
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 35
participants
  T790M mutation | 23
  MET amplification | 1
  SCLC Transformation | 3
  Unknown | 4
  Insufficient Tissue | 4

2. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically every 8 weeks on treatment (cycle duration=4 weeks). Participants were treated until evidence of disease progression or unacceptable toxicity. Progression follow-up was up to 3 years in this study cohort.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 60
months | 11.1 [9.1 to 14.8]

3. Post Hoc Outcome: Time to Repeat Biopsy
Description: Time to repeat biopsy is the duration of time from clinical determination of progressive disease to time of repeat biopsy.
Time Frame: At time of removal from study, patients were asked to undergo a repeat biopsy of their progressing or new tumor lesion. Progression follow up was up to 3 years in this study cohort.
Population: The analysis dataset is comprised of all evaluable patients.
Measure: Median (Full Range); unit: days
Arm/Group | Erlotinib
Number analyzed (Participants) | 35
days | 12 [0 to 97]

4. Post Hoc Outcome: Feasibility Rate
Description: Feasibility in this study is defined as the percentage of patients who completed a repeated biopsy per protocol after evidence of disease progression.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all patients eligible for repeat biopsy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 44
percentage of participants | 79.5 [67.0 to 88.9]

ADVERSE EVENTS:
Time Frame: Assessed each cycle on treatment up to day 30 post-treatment. Median (range) treatment duration for this study cohort was 10 months (1-62 months).
Description: Serious adverse events (AEs) per protocol are reported. For Other AEs, maximum grade toxicity by type (based on CTCAEv3 which includes coding events as 'Other') for a patient over time including only events with treatment-attribution of possibly, probably or definitely was calculated. A patient appears only once for a given type of toxicity. Patients with reports of multiple toxicities of different types are reported multiple times under the relevant toxicity categories.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 5/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=60)
Viral Enteritis (Gastrointestinal disorders) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Abdomen NOS (Infections and infestations) | 1
Hemorrhage, GI - Abdomen NOS (Gastrointestinal disorders) | 1
Ulcer, colon (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cardiac - ischemia (Cardiac disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac General-Other (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=60)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Infection Gr0-2 neut, conjunctiva (Infections and infestations) | 1
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, ungual (Infections and infestations) | 2
Infection w/ unk ANC conjunctiva (Infections and infestations) | 1
Infection w/ unk ANC mucosa (Infections and infestations) | 1
Infection w/ unk ANC oral cavity/gums (Infections and infestations) | 1
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Hematologic-other (Blood and lymphatic system disorders) | 5
Dry eye syndrome (Eye disorders) | 9
Eyelid dysfunction (Eye disorders) | 1
Ocular surface disease (Eye disorders) | 2
Tearing (Eye disorders) | 1
Ocular-other (Eye disorders) | 11
Chelitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 49
Distention/bloating, abdominal (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 4
Muco/stomatitis (symptom) esophagus (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 18
GI-other (Gastrointestinal disorders) | 4
Upper GI, hemorrhage NOS (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 2
Oral cavity, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 26
Fever w/o neutropenia (General disorders) | 1
Rigors/chills (General disorders) | 1
Edema limb (General disorders) | 2
Pain-other (General disorders) | 2
Syndromes-other (General disorders) | 1
Infection Gr0-2 neut, skin (Infections and infestations) | 3
Infection Gr0-2 neut, ungual (Infections and infestations) | 1
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 1
Infection w/ unk ANC vagina (Infections and infestations) | 2
Infection-other (Infections and infestations) | 2
Leukocytes (Investigations) | 3
Neutrophils (Investigations) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 9
Alkaline phosphatase (Investigations) | 5
ALT, SGPT (Investigations) | 8
AST, SGOT (Investigations) | 15
Bilirubin (Investigations) | 11
Metabolic/Laboratory-other (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 1
Taste disturbance (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 1
Neuropathy CN IX pharynx ear tongue (Nervous system disorders) | 1
Neuropathy CN XII tongue (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 1
Neuropathic, pain (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 36
Alopecia (Skin and subcutaneous tissue disorders) | 19
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 13
Pruritus/itching (Skin and subcutaneous tissue disorders) | 12
Rash/desquamation (Skin and subcutaneous tissue disorders) | 42
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 19
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Skin-other (Skin and subcutaneous tissue disorders) | 21
Scalp, pain (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Vascular-Other (Specify) (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No